CLINICAL TRIAL: NCT01315470
Title: Phase 1 Study of the Use of Granulocyte Colony-stimulating Factor for the Treatment of Repeated Implantation Failure in IVF Patients
Brief Title: Use of Granulocyte Colony-stimulating Factor for the Treatment of Recurrent Implantation Failure in IVF Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr Einat Zivi, organizational affiliation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCSF-HMO-CTIL
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Infertility
Keywords: improving pregnancy rate and endometrial thickness
MeSH Terms: conditions — Infertility | interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- neupogen (Experimental)
  Interventions: Drug: neupogen administration for women with recurrent IVF failure
- no intervantion (No Intervention)

INTERVENTIONS:
Drug: neupogen administration for women with recurrent IVF failure — neupogen 300 mcg - twice
  Other Names: GCSF injection; filgrastim
  Arms: neupogen

SUMMARY:
The investigators use granulocyte colony-stimulating factor (GCSF) for the treatment of recurrent implantation failure in IVF patient with cause unknown or due to thin endometrium. Several studies showed that GCSF improves embryo development and implantation and increase pregnancy rate.

DETAILED DESCRIPTION:
The investigators use granulocyte colony-stimulating factor (GCSF) for the treatment of repeated implantation failure (5 cycles) in IVF patient with cause unknown or due to thin endometrium. we intend to treat with GCSF during the IVF cycle if thin endometrium (<6 mm) is the cause for the treatment failure, and during the implantation window if cause unknown.

ELIGIBILITY:
Inclusion Criteria:

1. women after 5 failures in IVF cycles with cause unknown.
2. women after 5 failures in IVF due to thin endometrium (<6 mm) and unresponsive to estrogen supplements.

Exclusion Criteria:

1. history of hematology disease
2. allergy to GCSF
3. neutrophilia
4. severe lower back pain
5. liver dysfunction
6. hyperuricemia
7. a recent febrile disease or pneumonia
8. rheumatoid arthritis 9. sickle cell disease-

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-01 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate | 18 months

SECONDARY OUTCOMES:
endometrial thickness during IVF treatment | 18 months
endometrial thickness | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: einat zivi, MD, Principal Investigator
Locations (2):
- Israel (2):
  - Hadassah Ein Karem, Jerusalem, Israel
  - Hadassah Ein Karem, Jerusalem

REFERENCES:
- See also: 3. GM-CSF regulation of embryo development and pregnancy. Robertson SA. Cytokine Growth Factor Rev. 2007 Jun-Aug;18(3-4):287-98 — http://www.ncbi.nlm.nih.gov/pubmed/17512774